CLINICAL TRIAL: NCT04790097
Title: Safety and Preliminary Efficacy of Hipofractionated Irradiation Based on Dual FET-PET in Patients With Primary Glioblastoma Multiforme With Concomitant Temozolomide
Brief Title: FET-PET Directed Simultaneous In-field Boost for Primary GBM
Acronym: dualFETboost
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Franciszek Lukaszczyk Memorial Oncology Center (Other)
Responsible Party: Principal Investigator, Maciej Harat, M.D Ph.D., Prof. Franciszek Lukaszczyk Memorial Oncology Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FET-PET SIB Boost
Record Dates: First submitted 2021-01-23; First posted 2021-03-10 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Glioblastoma Multiforme
Keywords: FET-PET; Boost; Glioblastoma; Dose-intesification; Dose-escalation
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simultaneous In-Field Boost on FET-PET positive target volumes (Experimental)
  Interventions: Radiation: Moderately Hypofractionated Radiotherapy using Simultaneous In-Field Boost

INTERVENTIONS:
Radiation: Moderately Hypofractionated Radiotherapy using Simultaneous In-Field Boost — 78Gy in 30 fractions on FET-PET based target volumes;
  60Gy in 30 fractions on 2cm margin from MRI based target volumes;
  all patients will be treated with concomitant and adjuvant temozolomide

SUMMARY:
The combination of anatomical MRI examination with functional examination of tissue metabolic activity such as FET-PET (PET using the radiotracer - 18F-fluoro-ethyl-tyrosine) is a valuable tool to determine the actual tumor infiltration. The FET-PET examination can be performed using the dual-time point aqusition of FET for exact treatment planning. It has also been proven that using the dual FET-PET method, it is possible to obtain a precise image of the glioblastoma infiltration corresponding to the location and shape of the recurrence, and the tumor volumes in dual FET-PET are significantly larger than in MRI. Moreover, tumor defined in dual FET-PET is different than that of the tumor defined in single FET-PET acquisition.

In the DualFETboosT trial we plan to assess the safety and preliminary efficacy of hypofractionated irraditon using simultaneous in-field boost directed on dual FET-PET based tumor volumes for treatment of primary glioblastoma multiforme with concomitant temozolomide.

DETAILED DESCRIPTION:
In the case of the treatment of glioblastoma multiforme, as a standard, radiotherapy lasts 6 weeks, and the extension of treatment may adversely affect the tumor cells death, the patient's well-being and treatment costs (prolonged hospitalization). In turn, escalating the dose may increase the toxicity of radiation therapy by increasing DNA damage in healthy brain tissue. Using of dual FET-PET images for treatment planning allow to reduce volumes of healthy tissue irradiated. Dose-intensification proposed in the study using simultaneous in-field boost allows the dose escalation without increasing the overall treatment time. All patient will be treated with moderately hypofractionated radiotherapy (2.6 Gy per fraction) directed on PET positive volumes and conventional fractionation (60Gy in 30 fractions) on tumor margin.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological confirmation of glioblastoma (WHO grade IV)
* Age between 18-75 years of age
* General condition according to the Zubrod scale 0 or 2
* The results of the blood counts are normal
* Liver enzyme parameters normal
* The results of the parameters of the patient's functions are normal
* Informed consent to participate in the category

Exclusion Criteria:

* Coexistence of another cancer
* The location of the tumor in the area of the brain stem or cerebellum
* Prior brain radiation therapy
* No uptake visible in the FET-PET imaging
* Contraindications for MRI
* Contraindications to radiotherapy or chemotherapy
* Pregnancy, lack of consent to the use of protection against pregnancy, puerperium
* Alcohol addiction
* Mental illness
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | assessed up to 24 months
  From date of surgery until the date of death from any cause, percent of patient that are alive 1 and 2 years after surgery

SECONDARY OUTCOMES:
Progression Free Survival | up to 24 months
  from the date of surgery until progression of the disease or the date of death from any cause assessed
Objective response | up to 9 months
  according to Rano criteria; from the end of radiation therapy
Location of treatment failure | up to 24 months
  from the end of radiation therapy up to progression until progression of the disease or the date of death from any cause; according to irradiation field
Radiation necrosis | assessed up to 24 months
  from the end of radiation therapy up to progression until progression of the disease or the date of death from any cause; histopathological diagnosis of radiation necrosis
Side effects | up to 6 months
  from the end of radiation therapy up to progression until progression of the disease or the date of death from any cause; CTCAE grade 3 or higher

OTHER OUTCOMES:
FET predictive value | up to 24 months
  From date of surgery until the date of death from any cause, Correlation between FET uptake and survival

CONTACTS AND LOCATIONS:
Locations (1):
- The Franciszek Lukaszczyk Oncology Center, Bydgoszcz, Poland

REFERENCES:
- [Derived] Harat M, Blok M, Miechowicz I, Wiatrowska I, Makarewicz K, Malkowski B. Safety and Efficacy of Irradiation Boost Based on 18F-FET-PET in Patients with Newly Diagnosed Glioblastoma. Clin Cancer Res. 2022 Jul 15;28(14):3011-3020. doi: 10.1158/1078-0432.CCR-22-0171. PMID 35552391